CLINICAL TRIAL: NCT04879485
Title: Prehospital Plasma or Red Blood Cell Transfusion Strategy in Major Bleeding; PRIEST Trial
Brief Title: Prehospital Transfusion Strategy in Bleeding Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Norwegian Air Ambulance Foundation (Other); Odense University Hospital (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-289-20
Record Dates: First submitted 2021-04-29; First posted 2021-05-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Hemorrhage; Blood Component Transfusion
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard transfusion (No Intervention): Includes standard transfusion with a mixture of red blood cells and plasma
- Plasma (Active Comparator): Transfusion with plasma
  Interventions: Biological: Blood products
- Red Blood cells (Active Comparator): Transfusion with red blood cells
  Interventions: Biological: Blood products

INTERVENTIONS:
Biological: Blood products — Compare two different transfusion strategies against standard transfusion regimen
  Arms: Plasma; Red Blood cells

SUMMARY:
The aim of study is to compare clinical and biochemical effect of three different transfusion strategies among patients with major hemorrhage requiring prehospital transfusion.

A) Present prehospital standard treatment including a mixture of plasma and Red blood cell transfusion (RBC) transfusion B) Red blood cell transfusion (RBC) only C) Plasma transfusion only

Hypothesis:

1. Transfusion strategy including a mixture of RBC and plasma is superior as compared with only plasma or only RBC strategy in terms of initial treatment of circulatory shock (expressed as base deficit).
2. Endothelial function and ability of clot formation is preserved to a greater extent in patients receiving plasma.

DETAILED DESCRIPTION:
Rationale for the study:

The warranted clinical question to be unsolved is whether initial pre-hospital transfusion in bleeding patients should base on a strategy including plasma, RBC or combination of both.

Despite possible benefits, allogenic blood product are associated with side effects and pose significant logistic challenges in the prehospital environment. So far, a majority of the present knowledge is based on retrospective evaluations or clinical trials without relevant control groups.

ELIGIBILITY:
Inclusion Criteria:

* Major bleeding requiring prehospital transfusion

Exclusion Criteria:

* Transfusion with blood products already initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Base deficit | At hospital arrival (with in 1 hour)
  Arterial-gas analysis upon arrival with parameter base deficit as primary outcome

SECONDARY OUTCOMES:
30 days mortality | mortality within 30 days
  Mortality, follow up in patient records
Activated Partial Thromboplastin Time (APTT) | At hospital arrival (with in 2 hours)
  Plasma sample analysed; APTT
Endogenous thrombin potential (ETP) | At hospital arrival (with in 2 hours)
  Plasma sample analysed; thrombin generation assay
International Normalized Ratio (INR) | At hospital arrival (with in 2 hours)
  Plasma sample analysed; INR
Endothelium markers | At hospital arrival (with in 2 hours)
  Plasma sample analysed; Syndecan-1
Endothelium markers | At hospital arrival (with in 2 hours)
  Plasma sample analysed; soluble thrombomodulin
In hospital red blood cell transfusion requirements | Within in the first 24 hours after hospital arrival
  Amount of red blood cells transfused as registered in patient electronic records
In hospital plasma transfusion requirements | Within in the first 24 hours after hospital arrival
  Amount of plasma transfused as registered in patient electronic records
In hospital platelet transfusion requirements | Within in the first 24 hours after hospital arrival
  Amount of platelet transfused as registered in patient electronic records

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fenger-Eriksen, Study Chair — Aarhus Universityhospital
Locations (2):
- Denmark (2):
  - Aarhus Universityhospital, Silkeborg, Central Jutland
  - Danish Air Ambulance, Aarhus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066